CLINICAL TRIAL: NCT03790150
Title: National Approach to Standardize and Improve Mechanical Ventilation Care for Critically Ill Patients in Saudi Arabia
Brief Title: National Approach to Standardize and Improve Mechanical Ventilation
Acronym: NASAM
Status: Completed | Type: Observational
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Dr Yaseen Arabi, Chairman, Intensive Care Unit, King Abdullah International Medical Research Center
Other Study IDs: RC 17/223
Record Dates: First submitted 2018-12-20; First posted 2018-12-31 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Mechanical Ventilation Complication
Keywords: Ventilator-associated pneumonia; Mechanical Ventilation; Ventilator-associated events; Intensive care unit; Quality improvement project
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically Ventilated Patients: All patients admitted to the critical care unit and require mechanical ventilation
  Interventions: Other: Evidence-based practices

INTERVENTIONS:
Other: Evidence-based practices — Implementation of evidence-based practices

SUMMARY:
This is a pre-post implementation cohort study. This is a data driven quality improvement project which aims to improve the care of mechanically ventilated patients through the implementation of a bundle of evidence based practices, with a goal of reducing ventilator associated events and mortality.

DETAILED DESCRIPTION:
NASAM is a national collaborative quality improvement project in Saudi Arabia which aims to:

1. Reduce the rate of ventilator-associated events
2. Improve the compliance with NASAM bundle elements
3. Reduce the mortality of mechanically ventilated patients

The plan of this quality improvement project is to extend the implementation to a total of 100 ICUs in collaboration with multiple health systems across the country. A significant component of this project includes measuring the safety culture of ICUs.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to intensive care units

Exclusion Criteria:

* Age less than 14 years old

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mechanically ventilated patients
Sampling Method: Non-Probability Sample
Enrollment: 27966 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Ventilator-associated events | 18 months
  Ventilator-associated events rate per 1000 ventilator days in 18 months

SECONDARY OUTCOMES:
Sub-glottic endotracheal tube compliance rate | 18 months
  The percentage of ventilator days with sub-glottic endotracheal tube use
Head of bed elevation compliance rate | 18 months
  The percentage of ventilator days with head of bed elevation ≥30 degrees
Spontaneous awakening trial (SAT) compliance rate | 18 months
  The percentage of ventilator days with spontaneous awakening trial (SAT)
Percentage of ventilated patient days without sedation | 18 months
  The percentage of ventilated patient days without sedation use
Spontaneous breathing trials (SBT) compliance rate | 18 months
  The percentage of ventilator days with spontaneous breathing trial (SBT)
Percentage of ventilated patient days without neuromuscular blockers | 18 months
  The percentage of ventilated patient days without neuromuscular blockers
Percentage of out of bed mobility | 18 months
  The percentage of ventilated patient days with out of bed mobility
Percentage of CAM-ICU negative (no delirium) | 18 months
  The percentage of ventilator days with CAM-ICU negative (no delirium)
90-day mortality | 90 days
  The 90-day ICU mortality rate of ventilated patients
Mechanical ventilation duration | 90 days
  The duration of mechanical ventilation in calendar days
ICU length of stay | 90 days
  The number of calendar days from ICU admission to discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Yaseen M Arabi, MD, Principal Investigator — King Abdullah Medical City, Ministry of National Guard Health Affairs
Locations (2):
- Saudi Arabia (2):
  - Intensive Care Unit, King Abdulaziz Medical City, National Guard Health Affairs, Riyadh
  - King Abdullah International Medical Research Center, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arabi YM, Al Aseri Z, Alsaawi A, Al Khathaami AM, Al Qasim E, Alzahrani AA, Al Qarni M, Abdukahil SAI, Al-Dorzi HM, Alattasi A, Mandourah Y, Alaama TY, Alabdulaali MK, Alqahtani A, Shuaibi A, Al Qarni A, Alkatheri M, Al Hazme RH, Vishwakarma RK, Aldibasi O, Alshahrani MS, Attia A, Alharthy A, Mady A, Abdelrahman BA, Mhawish HA, Abdallah HA, Al-Hameed F, Alghamdi K, Alghamdi A, Almekhlafi GA, Qasim SAH, Al Haji HA, Al Mutairi M, Tashkandi N, Alabbasi SO, Al Shehri T, Moftah E, Kalantan B, Matroud A, Naidu B, Al Zayer S, Burrows V, Said Z, Soomro NA, Yousef MH, Fattouh AA, Tahoon MA, Muhammad M, Alruwili AM, Al Hanafi HA, Dandekar PB, Ibrahim K, AlHomsi M, Al Harbi AR, Saleem A, Masih E, Al Rashidi NM, Amanatullah AK, Al Mubarak J, Al Radwan AAA, Al Hassan A, Al Muoalad S, Alzahrani AA, Chalabi J, Qureshi A, Al Ansari M, Sallam H, Elhazmi A, Alkhaldi F, Malibary A, Ababtain A, Latif A, Berenholtz SM; Saudi Critical Care Trials Group. Impact of a national collaborative project to improve the care of mechanically ventilated patients. PLoS One. 2023 Jan 30;18(1):e0280744. doi: 10.1371/journal.pone.0280744. eCollection 2023. PMID 36716310